CLINICAL TRIAL: NCT01236508
Title: Relation of Carotid Artery Plaque Inflammation, Covert Stroke and White Matter Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulties recruiting this population for study population
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: The Ottawa Hospital (Other)
Responsible Party: Principal Investigator, Terrence Ruddy, Principal Investigator, Ottawa Heart Institute Research Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20100606-01H
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: TIA; Stroke; Carotid Artery Stenosis
Keywords: White Matter Hyperintensity; Stroke; Carotid Artery Plaque Inflammation; FDG PET; MRI; TIA
MeSH Terms: conditions — Stroke; Carotid Stenosis | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nuclear imaging (Experimental): PET/CT imaging with F-18 fluorodeoxyglucose
  Interventions: Radiation: PET/CT imaging with F-18 fluorodeoxyglucose

INTERVENTIONS:
Radiation: PET/CT imaging with F-18 fluorodeoxyglucose — Dose of 5 MBq/kg F-18-FDG given to fasting participant. Nuclear whole body imaging starting at 3 hours post-injection. The relation of the PET/CT image results and both the number of covert brain infarcts and the extent of white matter MRI hyperintensity will be investigated.

SUMMARY:
The investigators hypothesize that inflammation in carotid plaque is predictive of the extent of ischemic lesion burden on the brain and will add to risk stratification for individuals with carotid disease.

DETAILED DESCRIPTION:
Objectives:

1. To investigate the relationship of carotid inflammation, as measured by FDG positron emission tomography (PET) to standardized uptake value in atherosclerotic plaque, with the number of covert brain infarcts.
2. To investigate the relationship of FDG PET standardized uptake value with the relative volume of white matter hyperintensity.
3. To correlate vascular inflammation in the entire aorta and aortoiliac vessels to carotid inflammation and cerebral infarcts and white matter disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or greater at time of enrollment
* Written informed consent from patient or legal representative
* Diagnosis of stroke or TIA made by a stroke specialist within 90 days and fulfilling the following criteria:
* A TIA must involve a focal speech/language, motor or visual deficit (transient monocular blindness, amaurosis fugax) referable to the distribution of a carotid artery and lasting less than 24 hours.
* A stroke consisting of deficits as noted above with duration greater than 24 hours and/or confirmed on cerebral imaging. Post event Modified Rankin Score of 2 or less.
* Stroke meets the Trial of ORG 10172 in Acute Stroke Treatment (TOAST) criteria for large artery atherosclerosis
* Carotid Doppler, CTA or MRA confirming the presence of bilateral atherosclerotic disease resulting in carotid stenosis of any degree. Stenosis will be measured following the method used in NASCET for CTA and MRA. Carotid Doppler measurements will follow the criteria defined by the Society for Ultrasound consensus conference.
* 12 lead ECG or Holter monitor confirming the absence of atrial fibrillation.

Exclusion Criteria:

* TIA or stroke in the vertebrobasilar system
* Index event was primary hemorrhage
* History of intermittent atrial fibrillation
* Cardiac source of embolus suspected as cause of index event (artificial valve, segmental or global LV dysfunction, congenital cardiac defect)
* Diagnosis of vasculitis, dissection, or non-atherosclerotic carotid disease (Ehlers-Danlos, Marfans)
* Sinovenous thrombosis, endocarditis or hypercoagulable state
* Pacemaker, ICD or other contraindications to MRI
* Diminished Kidney Function
* Contraindication to radiation exposure (eg: pregnancy)
* Severe Claustrophobia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-11; Primary Completion 2016-10-27 (Actual); Study Completion 2016-10-27 (Actual)

PRIMARY OUTCOMES:
Plaque Inflammation | 30 days
  The extent to which plaque inflammation, as measured by the extent of FDG uptake, contributes to the number of covert infarcts and the magnitude of white matter hyperintensity.

CONTACTS AND LOCATIONS:
Overall Officials: Terrence Ruddy, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Civic Campus, Ottawa, Ontario, Canada